CLINICAL TRIAL: NCT06858774
Title: Use of Circadian Reset Technology to Alter REM Sleep and Appetitive Control Through Improved Network Connectivity in Brain in Patients With Binge Eating Disorder
Brief Title: Use of Circadian Reset Technology to Alter REM Sleep and Appetitive Control in Patients With Binge Eating Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Tom Hildebrandt, Professor and Chief of the Division of Eating & Weight Disorders, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY-24-01454
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Binge-Eating Disorder
Keywords: Binge Eating Disorder; Eating Disorder; Eating Disorder Treatment; Circadian Rhythm Technology; Virtual Reality
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: This is a Phase II clinical trial testing CRT in 20 individuals with Binge Eating Disorder to determine if this technology alters eating behavior and sleep quality using 10 minutes of daily exposure for 1 month.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will take place in this study to assign participants to the stimulation condition (getting CRT or control). The randomization module in REDCap will be used to perform randomization placement. The study staff and participants will be blind to condition. Only the project manager will know which headsets have CRT and which are control, all other staff will be blind to designation in REDCap. As the use procedures are equivalent, problem solving set up or use can be done by staff without breaking blind as the interface and use are equivalent in each condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circadian Reset Technology (Experimental): Participants will be given the headset to use for 5 minutes twice a day for 1 month while sitting in a resting position. Use will be separated by 12-16 hours of wakefulness.
  Interventions: Behavioral: Circadian Reset Technology
- VR Headset (Sham Comparator): Participants will be given a headset to use for 5 minutes twice a day for 1 month while sitting in a resting position. Use will be separated by 12-16 hours of wakefulness.
  Interventions: Behavioral: VR Headset

INTERVENTIONS:
Behavioral: Circadian Reset Technology — Circadian reset technology is a software used on a VR headset in this intervention. The software is a passive viewing experience like a guided meditation that presents visual images.
  Arms: Circadian Reset Technology
Behavioral: VR Headset — The software used on a VR headset in this intervention is a passive viewing experience like a guided meditation that presents neutral images that mimics the sequence used in the CRT software.
  Arms: VR Headset

SUMMARY:
This project includes testing circadian reset technology (CRT) on frequency of binge eating in a sample of 40 individuals with binge eating disorder. Participants will be randomized to one of two groups. Both groups use a virtual reality (VR) headset for 10 minutes (5 upon waking, 5 before sleep) daily for 1 month. One group will use the CRT software on the headset and the other group will use a software intended to be a control. Measures will be taken at baseline and 1-month. The researchers anticipate that use of CRT will improve sleep quality leading to increased appetitive control.

DETAILED DESCRIPTION:
This is a clinical trial with total of 40 individuals with Binge Eating Disorder ages 18 or older will be enrolled to use a VR headset with CRT or without. Examine whether 1-month of CRT alters binge eating frequency. Secondary outcomes include examining whether 1-month of CRT alters sleep quality, appetite regulation, functional magnetic resonance imaging (fMRI) measures of functional connectivity, food-based impulsivity/craving, and mood. Assessments are completed at baseline, weekly for 1 month, and then a final 1-month follow-up. Procedures include a screening/baseline phase to determine eligibility, gather baseline measures, and set-up on VR headset. Weeks 1 through 4 include using a VR headset twice a day for 5 minutes each. An online weekly survey will be completed, as well as daily ecological momentary assessment (EMA) surveys related to eating patterns throughout each day. The final visit will include a repeat of the baseline procedures including the fMRI. All recruitment and study procedures will take place through the Center of Excellence in Eating and Weight Disorders at the Icahn School of Medicine at Mount Sinai.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18+
* Diagnosed with Binge Eating Disorder using EDA-5
* English-speaking

Exclusion Criteria:

* Pregnancy
* Acute suicide risk/active suicidal ideation
* PSQI score <5 indicating good sleep quality
* A condition that may create a risk while using the VR headset including risk of falls, seizures, a heart condition, migraines, an eye or vision condition, or an inner ear condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in the total number of bulimic episodes | Baseline to 1-month
  Binge eating frequency measured by Eating Disorder Examination Questionnaire (EDE-Q). The EDE-Q scores behavioral features of eating disorders by calculating the number of episodes and number of days on which the behavior occurs. The total number of bulimic episodes will be measured to determine binge-eating frequency. Scores will be calculated between baseline and 1 month.
  The EDE-Q is a 28-item self-report measure assessing eating disorder symptoms. Full scale from 0-6, with higher score indicates greater severity of eating disorder symptoms.

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline to 1-month
  Sleep quality measured by Pittsburgh Sleep Quality Index (PSQI) is a 19-item assessment that measures sleep quality with questions about duration, latency, frequency/severity of sleep issues. Items are answered on a scale of 0-3. The final score is a total of all questions ranging from 0 to 21 with lower score indicating worse sleep quality and higher score indicating better sleep quality. Scores will be calculated between baseline and 1 month.
Change in Three-Factor Eating Questionnaire (TFEQ) | Baseline to 1-month
  Appetite regulation (restrained eating, disinhibited eating, and predisposition to hunger) measured by Three-Factor Eating Questionnaire (TFEQ) assesses appetite using 51 questions summarized in 3 subscales: cognitive restraint, uncontrolled eating, and emotional eating. Each item is scored as 0 or 1 and then summed. Subscales Cognitive restraint of eating score 0-21, Disinhibition score 0-16, and Hunger score 0-14. Full scale scored 0-51, higher scores indicate higher levels of restrained eating. Scores will be calculated between baseline and 1 month.
Changes in default mode network | Baseline to 1-month
  Change in Brain functional connectivity as measured by default mode network - This test measures the pattern of connectivity in the default mode network during rest. Strength of connectivity default mode network (DMN) will estimated at the network level and between individual nodes.
Change in Eating Loss of Control Scale (ELOCS) | Baseline to 1-month
  Food-based impulsivity measured by Eating Loss of Control Scale (ELOCS) measures the degree to which eating episodes included the feeling of loss of control measured continuously over the prior 4-weeks. There are 18 items scored on 0-10 scale from "not at all" to "Extremely/Completely". For total score, severity questions are averaged to get a mean severity score ranging between 0-10. Higher scores indicate more loss of control. Scores will be calculated between baseline and 1 month. Baseline to 1-month
Change in Food Cravings Questionnaire-Trait (FCQ-T) | Baseline to 1-month
  Food-based cravings (Trait) measure by Food Cravings Questionnaire-Trait (FCQ-T) is 39 items on a scale of 1 (never/NA) to 6 (always) with a total summed score ranging from 39 to 234 with higher scores indicating more frequent and intense food cravings. Scores will be calculated between baseline and 1 month.
Change in Food Cravings Questionnaire-State (FCQ-S) | Baseline to 1-month
  Food-based cravings (State) measured by Food Cravings Questionnaire-State (FCQ-S) has 15 items on a scale of 1 (strongly disagree) to 5 (strongly agree) with a total summed score ranging from 15 to 75 with higher scores indicating more intense food cravings. Scores will be calculated between baseline and 1 month.
Change in Depression Anxiety and Stress Scale (DASS) | Baseline to 1-month
  Depression Anxiety and Stress Scale (DASS) includes 42 questions that assess negative mood using subscales of depression, anxiety, and stress. Each subscale is scored 0-42, with total score from 0-126, higher score indicates poorer health outcomes.
  The depression scale scores are 0-9 (Normal), 10-13 (Mild), 14-20 (Moderate), 21-27 (Severe), and 28+ (Extremely Severe).
  The anxiety scale scores are 0-7 (Normal), 8-9 (Mild), 10-14 (Moderate), 15-19 (Severe), and 20+ (Extremely Severe).
  The stress scale scores are 0-14 (Normal), 15-18 (Mild), 19-25 (Moderate), 26-33 (Severe), and 34+ is (Extremely Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hildebrandt, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Department of Psychiatry, Eating and Weight Disorders Program, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared from this trial due to the early stages of investigation.